CLINICAL TRIAL: NCT04697888
Title: Use of Omegaven for Treatment With Parenteral Nutrition Associated Liver Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12010063
Record Dates: First submitted 2020-12-15; First posted 2021-01-06 (Actual); Results first posted 2021-03-12 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Parenteral Nutrition-related Hepatitis
MeSH Terms: interventions — fish oil triglycerides

STUDY DESIGN:
Intervention Model Description: This is a compassionate use protocol for patients with PNALD who have failed traditional treatment to receive Omegaven through an IND.

ARMS (1):
- Overall Study (Experimental): Use of Omegaven for patients with parenteral nutrition associated liver disease.
  Interventions: Drug: Omegaven

INTERVENTIONS:
Drug: Omegaven — Expanded Access Therapy with Omegaven will be initiated at a starting dose of 0.5 gm/kg/day to be infused over 24 hrs. After two days of infusion the dose will be increased to 1gm/kg/day.
  Other Names: IV Fish Oil Based Lipid Emulsion

SUMMARY:
To provide parenteral fat emulsion prepared from fish oil (omega-3 fatty acid emulsion, Omegaven®) to patients with liver disease (PNALD).

DETAILED DESCRIPTION:
This is a compassionate use protocol for patients with PNALD who have failed traditional treatment to receive Omegaven through an IND. Omegaven will be infused intravenously through either a central or peripheral catheter in conjunction with parenteral nutrition.

ELIGIBILITY:
Inclusion Criteria:

1. The patient will be PN dependent and unable to meet nutritional needs solely by enteral nutrition.
2. Patient will be <18 years of age.
3. Direct bilirubin > 2.0mg/dl
4. The patient must have failed standard therapies to prevent progression his/her liver disease.

Exclusion Criteria:

1. Other causes of chronic liver disease (Hepatitis C, Cystic fibrosis, biliary atresia, and alpha 1 anti-trypsin deficiency).
2. Patients who are allergic to eggs/shellfish
3. Patients who have severe hemorrhagic disorders.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel D Lim, MD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospitals and Clinics, Kansas City, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Overall Study
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Overall Study
Number analyzed (Participants) | 2
Age, Continuous [Mean (Standard Deviation); unit: Years] | 4.42 (3.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Disease Progression as Measured by Serum Levels of Hepatic Enzymes
Description: To evaluate whether established parenteral nutrition associated liver disease (PNALD) can be reversed or its progression halted by using a parenteral fat emulsion prepared from fish oil (omega-3 fatty acid emulsion, Omegaven®) as measured by normalization or decrease of serum levels of hepatic enzymes.
Time Frame: Up to 1 year
Population: No results recorded, study was utilized to provide compassionate use of study medication to participants.
Arm/Group | Overall Study
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Overall Study
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2012-01-30): https://cdn.clinicaltrials.gov/large-docs/88/NCT04697888/Prot_000.pdf